CLINICAL TRIAL: NCT02987387
Title: New Enrollment SAPIEN XT Post-Approval Study
Brief Title: COMPASSION XT PAS - Post-approval Study of the SAPIEN XT THV in Patients With Pulmonary Valve Dysfunction
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-10
Record Dates: First submitted 2016-10-19; First posted 2016-12-08 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis; Heart Defects, Congenital; Congenital Abnormalities; Cardiovascular Diseases; Heart Diseases
Keywords: Tetralogy of Fallot; Aortic Valve Defect/Disease Resulting in Ross Procedure; Transcatheter pulmonary valve implantation; Transcatheter pulmonary valve replacement; Pulmonary Atresia; Pulmonary Stenosis
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis; Heart Defects, Congenital; Congenital Abnormalities; Cardiovascular Diseases; Heart Diseases; Tetralogy of Fallot; Aortic Valve Disease; Pulmonary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TPVI: Transcatheter Pulmonary Valve Implantation with the SAPIEN XT THV
  Interventions: Device: SAPIEN XT THV

INTERVENTIONS:
Device: SAPIEN XT THV — SAPIEN XT THV will be implanted in the pulmonic position.

SUMMARY:
This study will confirm the safety and effectiveness of the Edwards Lifesciences SAPIEN XT Transcatheter Heart Valve (THV) System in patients with a dysfunctional right ventricular outflow tract (RVOT) conduit with a clinical indication for intervention in a post-market setting.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, multi-center clinical study to assess the safety and effectiveness of pulmonic implantation of the SAPIEN THV in patients with dysfunctional RVOT conduits requiring treatment for moderate or severe pulmonary regurgitation (PR) by transthoracic echocardiography (TTE) and/or RVOT conduit obstruction with a mean gradient of ≥ 35 mmHg by TTE.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a dysfunctional, non-compliant RVOT conduit.
2. The patient/patient's legally authorized representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Inability to tolerate an anticoagulation/antiplatelet regimen
2. Active bacterial endocarditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients with a dysfunctional, non-compliant right ventricular outflow tract (RVOT) conduit with a clinical indication for intervention.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Freedom from device- or procedure-related death or reintervention | 1 year

SECONDARY OUTCOMES:
Decrease in pulmonary regurgitation to mild or less for regurgitant lesions | 1 year
  Assessed via transthoracic echocardiogram (TTE)
Decrease in RVOT mean gradient to less than 30 mmHg for stenotic lesions | 1 year
  Assessed via TTE
Device Success | 48 Hours Prior to Discharge
  Device Success is a composite of:
  * Deployment of the valve to the target area, and
  * Removal of the delivery catheter out of the body, and
  * Improvement in pulmonary regurgitation to mild or less per the earliest evaluable TTE.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - The University of Iowa, Iowa City, Iowa
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Heart Center Nevada, Las Vegas, Nevada
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai Beth Israel, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No